CLINICAL TRIAL: NCT06665048
Title: Evaluating the Analgesic Efficacy of Oxycodone Hydrochloride in Pediatric Laparoscopic Cryptorchidism Surgery
Acronym: Anesthesia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shantou University Medical College (Other)
Responsible Party: Principal Investigator, Jiaxiang Chen, Shenzhen Children's Hospital, Shenzhen Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: szsetyyzjq@163.com
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Anesthesia; Oxycodone; Analgesia, Postoperative
Keywords: anesthesia; Oxycodone; Analgesia, postoperative
MeSH Terms: conditions — Agnosia | interventions — Oxycodone

STUDY DESIGN:
Intervention Model Description: Two-arm study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxycodone group (Experimental): Administer oxycodone hydrochloride (0.1 mg/kg) intravenously half an hour before surgery.
  Interventions: Drug: Oxycodone HCl
- Control group (No Intervention): The same routine anesthesia induction was given, and the same dose of normal saline was intravenously administered half an hour before the end of the operation to ensure that the operation conditions were the same as those of the control group except for the study drugs.

INTERVENTIONS:
Drug: Oxycodone HCl — Administer oxycodone hydrochloride (0.1 mg/kg) intravenously half an hour before surgery.
  Arms: Oxycodone group

SUMMARY:
Cryptorchidism surgery is a common pediatric procedure, often performed laparoscopically to reposition undescended testes into the scrotum. This technique involves manipulation and traction of the spermatic cord, which can lead to emergence agitation and short-term postoperative pain. Managing these symptoms effectively is essential for enhancing perioperative comfort and supporting faster recovery in children.

Oxycodone hydrochloride, a newer opioid with established analgesic effects in adult surgery, has been less studied in pediatric contexts. This randomized controlled trial aims to evaluate the effects of administering 0.1 mg/kg oxycodone hydrochloride 30 minutes before the end of laparoscopic cryptorchidism surgery in children aged 1 to 6. The study will assess outcomes such as anesthesia emergence time, extubation time, incidence of emergence agitation, postoperative analgesia, and nausea and vomiting. The goal is to determine if oxycodone hydrochloride could be an effective choice for pain relief in pediatric laparoscopic surgery, potentially reducing pain and complications, and providing clinical evidence to optimize anesthesia management for safer and more satisfactory pediatric surgical care.

This research aspires to contribute to the guidelines for pediatric anesthesia, offering a scientific basis for the clinical application of oxycodone hydrochloride in children.

DETAILED DESCRIPTION:
Oxycodone hydrochloride, a dual-opioid receptor agonist (μ and κ receptors), provides strong analgesic effects that can quickly alleviate intraoperative pain, enhancing pediatric patient comfort. It has a long duration of action, which supports sustained pain control during and after surgery, reducing the need for frequent dosing. In August 2015, the U.S. Food and Drug Administration (FDA) approved extended-release oxycodone for children with severe pain. Studies have shown that oral oxycodone has comparable pain relief to ibuprofen for children after fractures, highlighting its efficacy and safety profile. Compared to other analgesics, oxycodone hydrochloride has less impact on respiratory and circulatory systems, reducing perioperative risk and causing fewer side effects such as nausea and vomiting, aiding in smoother postoperative recovery.

A previous randomized, double-blind, parallel, multi-center trial demonstrated that intravenous patient-controlled oxycodone (0.1 mg/kg) provides effective postoperative pain relief for pediatric patients aged 3 months to 6 years undergoing elective surgery under general anesthesia, with a lower incidence of side effects than tramadol. However, research on its postoperative analgesic effects specifically in pediatric laparoscopic cryptorchidism surgery is limited, with insufficient data on hemodynamic stability during such procedures.

This study plans to administer intravenous oxycodone hydrochloride at 0.1 mg/kg 30 minutes before the end of surgery. Through a randomized controlled trial (RCT), we will evaluate oxycodone's effects on emergence agitation (assessed by PAED score), emergence and extubation times, postoperative pain (using the FLACC score), and postoperative nausea and vomiting (PONV score). The goal is to validate the efficacy of oxycodone hydrochloride in laparoscopic cryptorchidism surgery in children, providing evidence to support its rational clinical use.

Randomized controlled trial (RCT): The subjects were randomly divided into an experimental group (oxycodone hydrochloride group) and a control group (conventional anesthesia group) to compare the differences between the two groups.

Experimental group (O group): All children were fasted for 6 hours and 2 hours before surgery, and no preoperative medication was given. After the children woke up and entered the room, their heart rate (HR), non-invasive blood pressure monitoring (NIBP), pulse oximeter oxygen saturation (SpO2), respiratory rate (RR), and partial pressure of end-tidal carbon dioxide (PETCO2) were continuously monitored. Anesthesia induction was performed with 2-3 mg/kg propofol, 1 μg/kg remifentanil, and 0.4 mg/kg rocuronium intravenous injection, and the oxygen flow rate was 6 L/min. After the muscle relaxant took effect, a suitable laryngeal mask was inserted, and anesthesia was maintained with 2%-3% sevoflurane inhalation and remifentanil 0.2-0.4 μg/kg/min continuous pumping, and the oxygen flow rate was 2 L/min. Mechanical ventilation was performed using the tidal volume method, with a tidal volume of 6-8 mL/kg, a respiratory rate of 18-24 times/min, and an end-tidal carbon dioxide partial pressure of 30-35 mmHg. Hydroxycodone hydrochloride (0.1 mg/kg) was given intravenously half an hour before the end of the operation. Three minutes before the end of the operation, the oxygen flow was adjusted to 6 L/min, sevoflurane was discontinued, and the infusion of remifentanil was stopped. When the child's breathing was smooth and sufficient, and the spontaneous breathing tidal volume and frequency reached the extubation indication, the laryngeal mask was removed and sent to the PACU for further observation. When the child's Steward awakening score in the PACU was greater than 4 points, he was sent to the ward for continued monitoring of vital signs.

Control group (Group F): The same conventional anesthesia induction was given, and the same dose of normal saline was given intravenously half an hour before the end of the operation to ensure that the operation was the same as that of the control group except for the study drug.

Although oral oxycodone hydrochloride is widely used to relieve pediatric pain, few studies have explored intravenous administration for postoperative pain relief in children, and no research has yet reported its use in pediatric laparoscopic surgery. This study investigates the efficacy of intravenous oxycodone hydrochloride in preventing postoperative agitation, nausea, and vomiting, aiming to refine perioperative medication strategies for pediatric laparoscopic surgery and provide data to support precise clinical dosing.

The study employs a randomized, double-blind, controlled trial design with rigorous assessment methods to ensure reliability and validity of the findings. Postoperative agitation is evaluated using the PAED scale, with additional assessments for nausea and vomiting severity (PONV score) and pain (FLACC scale), creating a comprehensive, multidimensional evaluation system. This approach supports a thorough understanding of the drug combination's effects, providing a scientific basis for clinical decision-making.

Focused on pediatric cryptorchidism surgery, this study addresses a unique patient group, as infants and preschool children have specific anesthetic needs with heightened requirements for drug selection and dosing methods. By examining the safety and efficacy of oxycodone hydrochloride in this population, the research aims to offer new insights and methods for clinical anesthesia in pediatric laparoscopic surgery, supporting individualized treatment that enhances anesthetic efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Age range: patients between 1 and 6 years old who are scheduled to undergo cryptorchid surgery.
* No severe cardiopulmonary dysfunction, able to tolerate endotracheal intubation and general anesthesia.
* Children who have not received long-term analgesic medication before surgery.
* Children with a BMI range of 18.5-24 kg/m2.

Exclusion Criteria:

* History of allergy to oxycodone hydrochloride, fentanyl or other research-related drugs.
* Children who have severe pain or need long-term analgesic treatment.
* Combined with other serious diseases, such as malignant tumors, nervous system diseases, severe infections, coagulation disorders, congenital heart disease or other congenital malformations, and any other diseases that may interfere with the results of the study.
* Children who have received medication that may affect the evaluation of analgesic effects (such as other analgesics, sedatives, antidepressants, etc.) within two weeks before surgery.
* There are other situations that are not suitable for participation in this study, such as the child or family members cannot cooperate to complete the research requirements and may not be able to keep in touch during the study.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 162 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Emergence agitation | Within 30 minutes of emergencing
  The Pediatric Anesthesia Emergence Delirium (PAED) score is a standardized tool used to assess the presence and severity of emergence delirium (ED) in children following anesthesia. Emergence delirium is a post-anesthetic agitation or confusion commonly observed in young patients, characterized by behaviors such as crying, restlessness, and unresponsiveness. The PAED score evaluates these symptoms, helping clinicians gauge the need for interventions to manage postoperative agitation and ensure safe recovery.
  The PAED scale includes five behavioral items, each scored from 0 to 4, for a total score ranging from 0 to 20. A higher score indicates more severe agitation.

SECONDARY OUTCOMES:
Postoperative pain score | Within 30 minutes of emergencing
  The Face, Legs, Activity, Cry, Consolability (FLACC) score is a behavioral pain assessment tool commonly used to evaluate pain in children who are unable to communicate their pain verbally, including infants, young children, and those with cognitive impairments. The FLACC score is a reliable and widely used tool for assessing postoperative pain and discomfort in pediatric patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Children's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
Database not yet established

REFERENCES:
- [Background] Li S, Xiong H, Jia Y, Li Z, Chen Y, Zhong L, Liu F, Qu S, Du Z, Wang Y, Huang S, Zhao Y, Liu J, Jiang L. Oxycodone vs. tramadol in postoperative parent-controlled intravenous analgesia in children: a prospective, randomized, double-blinded, multiple-center clinical trial. BMC Anesthesiol. 2023 May 3;23(1):152. doi: 10.1186/s12871-023-02054-8. PMID 37138225
- [Background] Yang YT, Chen B, Bennett CL. FDA Approval of Extended-Release Oxycodone for Children With Severe Pain. Pediatrics. 2016 May;137(5):e20160205. doi: 10.1542/peds.2016-0205. Epub 2016 Apr 19. No abstract available. PMID 27244829
- [Background] Rohmah I, Chen YC, Lin CJ, Tsao NH, Chiu HY. Diagnostic accuracy of the pediatric CAM-ICU, pre-school CAM-ICU, Pediatric Anesthesia Emergence Delirium and Cornell Assessment of Pediatric Delirium for detecting delirium in the pediatric intensive care unit: A systematic review and meta-analysis. Intensive Crit Care Nurs. 2024 Jun;82:103606. doi: 10.1016/j.iccn.2023.103606. Epub 2023 Dec 29. PMID 38158251
- [Background] Wang Y, Chen L, Cui X, Zhou C, Zhou Q, Zhang Z. Clinical effect of minimally invasive surgery for inguinal cryptorchidism. BMC Surg. 2021 Jan 6;21(1):21. doi: 10.1186/s12893-020-01010-4. PMID 33407324